CLINICAL TRIAL: NCT03488303
Title: Impedance Pneumography Measurement During Acute Airway Obstruction and Recovery Phase in Young Children
Status: Completed | Type: Observational
Sponsor: Revenio Research (Industry)
Collaborators: Children's Hospital Srebrnjak (Other)
Responsible Party: Sponsor
Other Study IDs: VCS-006
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Obstruction; Airway, With Asthma
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main group: Study has only one group

SUMMARY:
The purpose of this study is to evaluate the association of signals recorded and analysed with Ventica® LFTS in infants and preschoolers during acute airway obstruction/asthma exacerbation and recovery thereof for changes in the IP-derived TBFV curves within and between nights.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-7
* Diagnosis of acute airway obstruction or asthma exacerbation requiring inpatient treatment

Exclusion Criteria:

* Need for an ICU treatment
* Bronchiolitis
* Pneumonia (not including viral infections)
* Other cardiorespiratory or neurological chronic diseases or states that may significantly alter the overnight breathing pattern
* Implanted or external active medical devices

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young children admitted to the ward at the hospital due to acute lower airway obstruction/asthma exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Association between clinical status and tidal breathing flow-volume (TBFV) curves | 2-4 nights while at ward
  Assess the association between clinical status and changes in tidal breathing flow-volume (TBFV) curves measured overnight with Ventica(R) Lung Function Testing System

SECONDARY OUTCOMES:
Association between lung function and tidal breathing flow-volume (TBFV) curves | 2-4 nights while at ward and 2 + 2 nights after discharge from hospital
  Assess the association between lung function (spirometry or oscillometry) and changes in tidal breathing flow-volume (TBFV) curves measured overnight with Ventica(R) Lung Function Testing System
Association between asthma control and tidal breathing flow-volume (TBFV) curves | 2 + 2 nights after discharge from hospital
  Assess the association between asthma control (C-ACT questionnaire) and changes in tidal breathing flow-volume (TBFV) curves measured overnight with Ventica(R) Lung Function Testing System

CONTACTS AND LOCATIONS:
Overall Officials: Davor Plavec, MD, PhD, Principal Investigator — Children's Hospital Srebrnjak
Locations (1):
- Children's Hospital Srebrnjak, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No